CLINICAL TRIAL: NCT07100249
Title: A Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of HDM2012 in Subjects With Advanced Solid Tumors
Brief Title: A Study of HDM2012 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HDM2012-101
Record Dates: First submitted 2025-07-16; First posted 2025-08-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HDM2012 (Experimental): In dose escalation phase, participants will be administered escalating doses of HDM2012 at 1.0~5.2mg/kg IV on Day 1 of repeated 21-day cycles. In dose expansion phase, participants will be administered to recommended dose for expansion (RDE) of HDM2012 on Day 1 of repeated 21-day cycles .
  Interventions: Drug: HDM2012

INTERVENTIONS:
Drug: HDM2012 — HDM2012 will be administered via IV infusion.

SUMMARY:
This is a first-in-human (FIH) study to evaluate the safety and preliminary efficacy of experimental drug HDM2012 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The participants understand and voluntarily (or their legally authorized guardian) sign a written informed consent form (ICF) approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC).
2. Males or females aged ≥18 years and less than or equal to 75 years.
3. For escalation cohorts in the dose escalation phase: subjects must have histologically or cytologically confirmed advanced or metastatic malignant solid tumors, who have been previously treated and failed after adequate standard therapy, and have no standard treatment options available that have the potential to confer clinical benefit, including but not limited to gastric cancer (including esophagogastric junction adenocarcinoma), colorectal cancer, pancreatic cancer, etc.
4. For backfill cohorts in the dose escalation phase and the dose expansion phase: subjects must have histologically or cytologically confirmed advanced or metastatic gastric cancer (including gastroesophageal junction adenocarcinoma) or colorectal cancer.
5. Tumor tissue samples must be sent to the central laboratory for immunohistochemical testing.
6. ECOG performance status of 0 - 1.
7. Expected survival time >3 months.
8. Per RECIST v1.1 criteria: Ia phase subjects in dose escalation cohort must have at least one evaluable lesion; Ia phase subjects in backfill cohort and Ib phase subjects must have at least one measurable lesion (tumor lesions in previously irradiated areas are not considered measurable unless clear radiographic progression post-radiation is documented; measurable lesions in Ib phase should exclude biopsy sites).
9. Adequate organ function demonstrated by screening laboratory tests (no growth factors or corrective treatments allowed within 14 days prior to screening tests).
10. Willingness of women of reproductive potential to observe conventional and highly effective birth control methods with failure rates of <1% for the duration of treatment and for 7 months following the last dose of study treatment; Willingness of men of reproductive potential to observe conventional and highly effective birth control methods with failure rates of <1% for the duration of treatment and for 4 months following the last dose of study treatment; this must include barrier methods such as condom or diaphragm with spermicidal gel. Women of reproductive potential have a negative serum pregnancy test within 7 days before study enrollment; For male participants with a nonpregnant female partner of child-bearing potential and a woman of child-bearing potential, one of the following highly effective birth control methods with a failure rate of less than 1% per year when used consistently and correctly are recommended .
11. Willing and able to complete scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Prior treatment with antibody-drug conjugates (ADCs) containing topoisomerase I inhibitors.
2. Subjects who have received the following treatments:

   1. Major surgery within 4 weeks prior to first dose, except minor procedures such as appendectomy, tumor biopsy, etc.;
   2. Radiation therapy to bone marrow (equivalent to pelvic marrow area) or extensive radiation within 4 weeks prior to first dose; local radiotherapy (e.g., thoracic vertebrae and rib radiation) within 2 weeks prior to first dose;
   3. Continuous systemic corticosteroid administration (>10 mg/day prednisone equivalent) within 2 weeks prior to first dose; low-dose corticosteroids (≤10 mg/day prednisone equivalent) are permitted if dose has been stable for 4 weeks;
   4. Subjects who have received other systemic anti-tumor therapies within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose, unless a scientifically justified washout period is provided, such as relevant PK/PD of the prior therapy and relevant clinical and laboratory parameters, based on the characteristics of preceding therapy.
3. Active malignancies within past 2 years, except studied cancer and cured localized tumors (e.g., basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ).
4. Subjects have not recovered from prior treatment-related or other anti-cancer therapy-related AEs (alopecia, ≤Grade 2 sensory neuropathy, or other ≤Grade 2 AEs deemed non-safety risks by investigator are acceptable) to ≤Grade 1 or baseline.
5. Known active central nervous system metastases. Untreated asymptomatic or treated brain metastasis subjects with radiologically confirmed stable status for ≥4 weeks and no need for steroids/antiepileptics ≥2 weeks may be enrolled. Leptomeningeal metastases (symptomatic or asymptomatic) must be excluded.
6. Subjects with any cardiovascular/cerebrovascular diseases/conditions/indications.
7. At screening, participants with active syphilis, immunodeficiency disease (HIV), active hepatitis (HBV, HCV), except for asymptomatic chronic hepatitis B or C carriers.
8. History of interstitial pneumonia, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia found on chest computed tomography (CT) during screening; previous use of hormone shock therapy for pneumonia.
9. Complete or incomplete intestinal obstruction or imaging findings indicating risk of intestinal obstruction.
10. Presence of other diseases that may affect the efficacy and safety of the IMP.
11. Presence of large or symptomatic moderate pleural effusion, pericardial effusion, or ascites during screening that remains poorly controlled despite treatments like drainage.
12. Unstable thrombotic events requiring therapeutic intervention within 6 months prior to screening, including deep vein thrombosis, arterial thrombosis, and pulmonary embolism; excluding catheter-related thrombosis.
13. Previous solid organ transplantation.
14. Known or suspected allergy to IMP components or their analogs.
15. Pregnant or breastfeeding women.
16. Investigator's judgment that the subject is unsuitable for participation (e.g., non-optimal treatment benefit, poor compliance, etc.).
17. Received strong or moderate CYP3A4 inhibitors or inducers within 1 week prior to dosing or 5 half-lives (whichever is longer), or anticipated need for long-term use of strong or moderate CYP3A4 inhibitors or inducers during study intervention and within 30 days after last dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events (for dose escalation phase) | up to 21 days following first dose
  DLT will be determined by definition during the DLT observation period.
Incidence and severity of adverse events(for dose escalation phase) | Until 30 days after the last dose or initiation of a new antineoplastic therapy, whichever occurs first
  The safety profile of HDM2012 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Objective Response Rate (ORR) (for dose expansion phase) | through study completion, an average of 1 year
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Recommended Phase 2 Dose (RP2D) (for dose expansion phase) | through study completion, an average of 1 year
  The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic, E-R relationships, and efficacy data.

SECONDARY OUTCOMES:
Plasma concentration of HDM2012 | up to7 days following last dose
  Plasma concentration of HDM2012
Immunogenicity | up to 7 days following last dose
  Number and percentage of anti-drug antibody (ADA)-positive patients will be assessed.
Incidence and severity of adverse events(for dose expansion phase) | Until 30 days after the last dose or initiation of a new antineoplastic therapy, whichever occurs first
  The safety profile of HDM2012 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Objective Response Rate (ORR)(for dose escalation phase) | through study completion, an average of 1 year
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Time to Response (TTR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  TTR is defined as the interval from the start of study therapy to the first documentation of an objective response.
Progression free survival (PFS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS is defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression/relapse or death from any cause.
Duration of Response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to100 months
  DOR is defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression/relapse or death from any cause.
Overall survival (OS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  OS is defined as the interval from the start of study therapy to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China